CLINICAL TRIAL: NCT00421395
Title: Phase I/II Radioimmunotherapy of Non-Hodgkin's Lymphoma With Radiolabeled Humanized IMMU-LL2: Treatment With 90Y-hLL2 IgG
Brief Title: Safety Study of NHL With 90Y-hLL2 IgG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: William Wegener, MD, PhD, Immunomedics, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL2-06EU
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2008-01

CONDITIONS: NHL; B-cell NHL; Non-Hodgkins Lymphoma
Keywords: NHL; B-cell NHL; Non-Hodgkins lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- multi (Experimental): escalating in increments of 2.5 mCi/m2
  Interventions: Biological: 90Y-hLL2

INTERVENTIONS:
Biological: 90Y-hLL2 — weekly dosing for either 2 or 3 weeks
  Other Names: epratuzumab; hLL2

SUMMARY:
This will be an open label, multiple center, non-randomized, dose-escalation Phase I/II trial, designed to evaluate the safety and effectiveness of a repeated, outpatient regimen utilizing IMMU-hLL2 intact monoclonal antibody IgG labeled with different doses of 90Y for the treatment of patients B-cell lymphoma (NHL).

DETAILED DESCRIPTION:
90Y-labeled hLL2 will be administered according to a schedule based upon whether or not a patient had prior high-dose chemotherapy with a marrow or stem cell transplant. Patients with both indolent and aggressive types of NHL will be enrolled at each dose level without segregation. However, at the conclusion of the trial, with the maximum tolerated dose (MTD) defined, a minimum number of 6 patients with indolent NHL, 6 patients with aggressive NHL, and 6 patients with >25% bone marrow involvement will be studied at that dose level.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologic or cytological diagnosis of B-cell lymphoma, and have failed at least one regimen of standard chemotherapy. All histologic grades of non-Hodgkin's lymphoma (NHL) will be eligible for these studies.
* Patients must be > 18 years of age
* Measurable disease by CT, with at least one lesion > 1.5 cm in one or both dimensions
* less than 25% bone marrow involvement as determined by bone marrow biopsy
* Patient must have greater than 15% cellularity of the bone marrow.
* Patients must be at least 4 weeks beyond any major surgery.
* Patients must be at least 4 weeks beyond any radiation therapy to the index lesion and must have recovered from radiation induced toxicity.
* Patients must be at least 4 weeks beyond prior chemotherapy and/or immunotherapy, or 2-weeks after corticosteroids, and their blood counts must be within the eligibility criteria. Corticosteroids may, however, be given concomitantly if used to treat adrenal insufficiency
* Patients must have a performance status of 70 or greater on the Karnofsky scale equivalent to ECOG 0-1 (See Appendix A) and a minimal life expectancy of 6 months.
* Patients must be able to give cognizant informed consent.

Exclusion Criteria:

* Patients with a significant concurrent medical complication including severe anorexia, nausea or vomiting that in the judgement of the Investigator could affect the patient's ability to tolerate or complete this study.
* Patients with metastasis to the brain.
* Patients with extensive irradiation to more than 25% of their red marrow will be excluded, except those who had total body irradiation in the context of bone marrow or stem cell transplantation regimen with subsequent engraftment of a functional marrow (i.e., resulting in normal peripheral blood counts). Subjects who have received external radiation to specific organs or areas at the maximum tolerated level are also excluded.
* Women who test positive for pregnancy.
* Patients with splenomegaly.
* Patients with > 4 treatment regimens prior to this protocol, including chemotherapy, radiotherapy and/or other immunotherapy.
* Patients with prior radioimmunotherapy treatments (unless for retreatment under this protocol).
* Patients receiving rituximab within 3 months, unless progressing after treatment.
* Patients with <50% LVEF by required MUGA or 2-D ECHO.
* Patients with <60% of predicted value by required pulmonary function tests.
* Patients who have active Hepatitis B or C or are known HIV positive.
* Patients with another primary malignancy (except basal/squamous cell carcinoma of the skin or carcinoma in-situ of the cervix.
* Patients with other serious medical, surgical, or psychiatric history, unless currently stable and well controlled, without significant increase in treatment medications for at least 30 days preceding study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2002-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated from physical examinations, hematology and chemistry testing and toxicity evaluation | First 12 weeks, total 5 years

SECONDARY OUTCOMES:
Determine maximum tolerated dose (MTD) | first 12 weeks
Evaluate the immunogenicity and safety of repeated infusions of 90Y-hLL2 in NHL patients. | 6 weeks, 12 weeks, every 3 months if HAHA elevated
Determine the therapeutic effects, in terms of objective response rate and duration, of the therapeutic agent in NHL patients. | 6 wks, 12 wks, every 3 mos for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William A Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (5):
- France (2):
  - Research Unit 463 INSERM, Nantes, Cedex
  - Service des Maladies du Sang, Lille
- Germany (3):
  - University Hospital Dresden, Dresden
  - Klinikum der Georg-August-Universitat Gottingen, Göttingen
  - Universitatsklinikum University of Saarland, Homburg/Saar

REFERENCES:
- [Background] Linden O, Hindorf C, Cavallin-Stahl E, Wegener WA, Goldenberg DM, Horne H, Ohlsson T, Stenberg L, Strand SE, Tennvall J. Dose-fractionated radioimmunotherapy in non-Hodgkin's lymphoma using DOTA-conjugated, 90Y-radiolabeled, humanized anti-CD22 monoclonal antibody, epratuzumab. Clin Cancer Res. 2005 Jul 15;11(14):5215-22. doi: 10.1158/1078-0432.CCR-05-0172. PMID 16033839
- [Background] Linden O, Tennvall J, Cavallin-Stahl E, Darte L, Garkavij M, Lindner KJ, Ljungberg M, Ohlsson T, Sjogreen K, Wingardh K, Strand SE. Radioimmunotherapy using 131I-labeled anti-CD22 monoclonal antibody (LL2) in patients with previously treated B-cell lymphomas. Clin Cancer Res. 1999 Oct;5(10 Suppl):3287s-3291s. PMID 10541377
- [Background] Hindorf C, Linden O, Stenberg L, Tennvall J, Strand SE. Change in tumor-absorbed dose due to decrease in mass during fractionated radioimmunotherapy in lymphoma patients. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):4003S-6S. PMID 14506200
- [Background] Sharkey RM, Burton J, Goldenberg DM. Radioimmunotherapy of non-Hodgkin's lymphoma: a critical appraisal. Expert Rev Clin Immunol. 2005 May;1(1):47-62. doi: 10.1586/1744666X.1.1.47. PMID 20477654
- [Background] Sharkey RM, Brenner A, Burton J, Hajjar G, Toder SP, Alavi A, Matthies A, Tsai DE, Schuster SJ, Stadtmauer EA, Czuczman MS, Lamonica D, Kraeber-Bodere F, Mahe B, Chatal JF, Rogatko A, Mardirrosian G, Goldenberg DM. Radioimmunotherapy of non-Hodgkin's lymphoma with 90Y-DOTA humanized anti-CD22 IgG (90Y-Epratuzumab): do tumor targeting and dosimetry predict therapeutic response? J Nucl Med. 2003 Dec;44(12):2000-18. PMID 14660727
- [Background] Griffiths GL, Govindan SV, Sharkey RM, Fisher DR, Goldenberg DM. 90Y-DOTA-hLL2: an agent for radioimmunotherapy of non-Hodgkin's lymphoma. J Nucl Med. 2003 Jan;44(1):77-84. PMID 12515879
- [Background] Lindén O, et al. Outcome and absorbed dose following 90-yttrium-epratuzumab in B-cell lymphoma, using a dose-fractionation schedule. (Abstract No. 1479) Blood 2003; 102/11:407a.
- [Background] Postema EJ, Borjesson PK, Buijs WC, Roos JC, Marres HA, Boerman OC, de Bree R, Lang M, Munzert G, van Dongen GA, Oyen WJ. Dosimetric analysis of radioimmunotherapy with 186Re-labeled bivatuzumab in patients with head and neck cancer. J Nucl Med. 2003 Oct;44(10):1690-9. PMID 14530488
- [Background] Leonard JP, Siegel JA, Goldsmith SJ. Comparative physical and pharmacologic characteristics of iodine-131 and yttrium-90: implications for radioimmunotherapy for patients with non-Hodgkin's lymphoma. Cancer Invest. 2003 Apr;21(2):241-52. doi: 10.1081/cnv-120016421. PMID 12743990
- [Background] Lindén O, et al. Radioimmunotherapy with Y-90-Epratuzumab in patients with previously treated B-cell lymphoma. A fractionated dose-escalation study. (Abstract 5.05 Hematology) Special Issue: World Congress of Nuclear Medicine, September 2002; 5/17.
- [Background] Liu, Huaitian, et al. Targeting the CD22 receptor with RNA damaging agents. Cancer Drug Discovery and Development: Tumor Targeting in Cancer Therapy. Edited by: M Pagé, Humana Press Inc., Totowa, NJ: 109-118
- [Background] Lindén O, et al. Durable response to 90-yttrium-epratuzumab (hLL2) in B-cell lymphoma failing chemotherapy by using dose-fractionation schedule. (Abstract presented at the American Society of Hematology 43rd Annual Meeting) Blood 2001; 98/11: 602a
- [Background] Hajjar G. et al. Phase I/II radioimmunotherapy trial with 90Y-labeled epratuzumab (LymphoCide; anti-CD22 monoclonal antibody) in relapsed/refractory non-Hodgkin's lymphoma (NHL). (Abstract #583) J Nucl Med Suppl, May 2001; 42/5: 156P.
- [Background] Goldenberg DM. The role of radiolabeled antibodies in the treatment of non-Hodgkin's lymphoma: the coming of age of radioimmunotherapy. Crit Rev Oncol Hematol. 2001 Jul-Aug;39(1-2):195-201. doi: 10.1016/s1040-8428(01)00108-1. PMID 11418316
- [Background] Juweid M, Schuster SL, et al. Updated results of radioimmunotherapy of relapsed/refractory non-Hodgkin's lymphoma with conventional and stem cell supported doses of 90Y-labeled humanized LL2 anti-CD22 monoclonal antibody. (Abstract #40) Cancer Biother & Radiopharm 2000, 15/4: 408
- [Background] Lindén O, Tennvall J, et al. A Phase I/II trial with Y-90 hLL2 in recurrent B-cell lymphomas. Preliminary results. (Abstract #67) Cancer Biother & Radiopharm 2000, 15/4: 413
- [Result] Bodet-Milin C, et al. FDG-PET predicts response to fractionated radioimmunotherapy with 90Y-epratuzumab anti-CD22 MAb in patients with NHL. (Abstract #4782) Blood 2995; 106/11:275b.
- [Result] Bodet-Milin C, et al. Positron emission tomography with F-18-fluorodeoxyglucose (PET-FDG) predicts response to fractionated radioimmunotherapy (RIT) using 90Y-epratuzumab in non-Hodgkin's lymphoma (NHL). (Abstract #1234) J Nucl Med Abstract Bk Suppl 2 2005; 46/5:379P.
- [Result] Chatal J-F, et al. Fractionated radioimmunotherapy in NHL with DOTA-conjugated humanized anti-CD22 epratuzumab at high cumulative 90Y doses. (Abstract #447) J Nucl Med Abstract Bk Suppl 2 2005; 46/5:155P.
- [Result] Chatal J-F, et al. Radioimmunotherapy in non-Hodgkin's lymphoma (NHL) using a fractionated schedule of DOTA-conjugated, 90Y-radiolabeled, humanized anti-CD22 monoclonal antibody, epratuzumab. (Abstract #2545) Proceedings of ASCO 2004; 23:174.
- See also: Related Info — http://www.immunomedics.com
- See also: Related Info — http://www.lrfa.org